CLINICAL TRIAL: NCT04072757
Title: Fruit and Vegetable Prescription Program
Acronym: FVRx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BETH COMERFORD (Other)
Responsible Party: Sponsor-Investigator, BETH COMERFORD, PRINCIPAL INVESTIGATOR, Griffin Hospital
Organization: Griffin Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-02
Record Dates: First submitted 2017-11-01; First posted 2019-08-28 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): The cooking skill building/nutrition education workshops will be led by a multidisciplinary team comprised of: a chef/instructor, a nutritionist and/or registered dietitian, MD and/or Preventive Medicine Resident, and Yale-Griffin Prevention Research Center staff. The cooking/nutrition education workshop sessions will be approximately 45 minutes and will: include a plant forward approach to healthy eating; integrate nutrition and health-related information and cooking instruction (i.e. knife skills, equipment use); show participants how to prepare meals that are simple, nutritious, affordable, and delicious; provide recipes and nutrition information aimed at improving dietary intake and health status; and provide an enjoyable program that participants will look forward to attending. Fruit and vegetable prescription vouchers will be redeemed at ShopRite grocery stores (Ansonia and Shelton locations) and Griffin Hospital's farmers market, where redemption will be tracked.
  Interventions: Behavioral: Intervention Group
- Control Group (Placebo Comparator): The control group will not receive vouchers or nutrition education/skill building but will be exposed to any standard Griffin Hospital worksite offerings. A "mini program" (2 -4 hours) workshop will be offered to participants in the control group, and all intervention materials will be provided.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Intervention Group — Session One: Loving Food That Loves You Back - Food as Fuel
  * connection nutrition and health Session Two: Myth busting: Fruits and Vegetables - delicious and affordable
  * seasonal fruits & vegetables in the diet Session Three: No Time to Cook! Making nutritious meals that are fast and easy
  * quickly make delicious/nutritious meals using minimal ingredients Session Four: Don't Eat Food You Can't Pronounce Except Quinoa; Eat Quinoa
  * choose healthier foods Session Five: Taste Bud Rehab
  * reduce foods high in sugar and salt.Mind-body connection Session Six: Batch & One Ingredient Cooking
  * making large quantities to freeze; one ingredient cooking Session Seven: Sweet Tooth? Healthy Desserts
  * prepare healthier desserts Session Eight: Family Meal Practices
  * healthy eating habits in children Session Nine: Snacks as Mini Meals
  * make nutritious snacks to keep energy up all day Session Ten: Revamp Your Favorite Recipe
  * "healthy up" favorite recipes
  Arms: Intervention Group
Behavioral: Control Group — The control group will not receive vouchers or nutrition education/skill building but will be exposed to any standard Griffin Hospital worksite offerings. A "mini program" (2 -4 hours) workshop will be offered to participants in the control group, and all intervention materials will be provided.
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine the effectiveness of a worksite based Fruit & Vegetable Prescription (Rx) Program designed to increase fruit and vegetable consumption and improve diet quality and other health outcomes of participants. The program includes incentives (coupons) and skill building/educational sessions to increase intake of fruits, vegetables, and other health promoting foods (i.e. legumes, whole grains). The program will focus on delicious, nutritious, affordable, simple and quick meal preparation.

DETAILED DESCRIPTION:
Hypotheses

* The program will increase intake of fruits, vegetables and other health promoting foods, and will improve diet quality.
* The program will improve household meal practices.
* The program will improve BMI, waist circumference, lipid panel, HbA1c, and blood pressure.
* Improvements in outcome measures will be sustained 3 months post intervention.

Specific Aims

* To determine the effect of a worksite based F&V Rx program as compared to control/no intervention on diet quality.
* To determine the effects of a worksite based F&V Rx program as compared to control/no intervention on household meal practices.
* To determine the effects of a worksite based F&V Rx program as compared to control/no intervention on BMI, waist circumference, lipid panel, HbA1c, and blood pressure.
* To determine whether improvements resulting from the program are sustainable over time.

Background In 2011-2012, two-thirds of adults and over 30% of children and adolescents in the U.S. were overweight or obese. Obesity is widely recognized as a grave public health concern because of its association with increased risk for a multitude of chronic diseases and other adverse health outcomes. The persistence of high obesity rates in children and adults in the U.S. and the low rates of adherence to current recommendations for fruit and vegetable consumption are evidence of the inadequacy of efforts to date to promote healthy lifestyles.

Adults-specifically, parents-have a strong influence on children's eating and physical activity habits. Children have innate preferences for sweet, energy-dense foods; however, some food preferences are learned. Early introduction and repeated exposure to healthy foods may help to familiarize and increase acceptance and liking of those foods. Parents can help children learn healthy eating habits by using appropriate child feeding practices, modeling the desired behaviors, and creating a home food environment that is conducive to healthy eating. Likewise, parents' physical activity behaviors may also influence children's activity levels. To achieve meaningful change in childhood obesity, it is necessary to change the culture of the entire household by reaching both adults and children.

Whereas children are often exposed to health promotion programming in schools, adults may be exposed to similar messages at work. There is an extensive literature on the capacity of worksites to effectively promote healthy lifestyles while reducing medical costs and absenteeism. Worksite interventions targeting fruit and vegetable consumption have been found to be effective, particularly when they include a focus on employees' families. Interventions that include a subsidy or financial incentive to reduce the cost of fruits, vegetables, and other healthy foods have also been shown to increase the purchase and consumption of those foods. However, there are few if any studies evaluating the effectiveness of a worksite-based intervention including financial incentives for fruit and vegetable purchases, nutrition education, and a focus on changing the behavior of the whole family.

ELIGIBILITY:
Inclusion Criteria:

1. Griffin employees, aged 18 and over, with a child/children enrolled in VITAHLS schools (Shelton, Ansonia, Derby, Seymour, and Naugatuck) - grades pre-k thru 12.
2. be able to attend weekly 45 minutes nutrition/cooking workshops.

Exclusion Criteria:

1. Inability to attend majority of the Nutrition and cooking workshops
2. Anticipated inability to complete study protocol for any reason
3. Diagnosis of cancer except skin cancer of less than 5 years or unstable treatment for less than 5 years.
4. Unstable angina or other significant cardiovascular condition, prior or planned bariatric surgery.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Diet quality | Up to 3 Months
  Participants will complete three 24-hour recalls using the web-based ASA24 - http://riskfactor.cancer.gov/tools/instruments/asa24/ (Automated Self-Administered 24-Hour Recall) at each of the 3 assessment time points (9 total). Diet quality will be assessed using the Healthy Eating Index 2010. The Prevention Research Center will have computers available for participants who do not have access to computers to complete the ASA24.

SECONDARY OUTCOMES:
Change in Household meal practices | Up to 3 Months
  The Meals in Our Household questionnaire will be used to assess changes in household meal practices (e.g. preparation, timing and location of meals; child behavior during meals, etc.). Because this instrument was designed for families with children between the ages of 3 and 11, it will only be administered to participants with children within this age range.
Change in Body Mass Index (BMI) | Up to 3 Months
  Body mass index (BMI) will be calculated as weight (kg) divided by height in meters (m) squared.
Change in Body Composition- Body Fat and Body Water Percentage | Up to 3 Months
  Body composition (Body Fat and Body Water Percentage) will be measured using bioelectrical impedance analysis, which uses the resistance of electrical flow through the body to estimate body fat and water. The Tanita SC-240 Body Composition Analyzer will be used to measure body composition. The SC-240 calculates body fat% and total body water%.
Change in Waist circumference | Up to 3 Months
  Waist circumference will be measured using the U.S. government standard protocol. To measure the waist circumference, the clinical research coordinator will ask the participant to stand and he/she will place a tape measure around the participant's middle, just above her/his hipbones, at the level of the belly button. The clinical research coordinator will ensure that the tape is horizontal around the participant's waist, and will then keep the tape snug around the participant's waist while not compressing the skin, and will measure her/his waist just after exhaling.
Change in Serum Lipids and HbA1c | Up to 3 Months
  Total cholesterol (Tchol), triglycerides (TG), and high-density lipoprotein (HDL) will be obtained by direct measurements. Very-low-density lipoprotein (VLDL) and low-density-lipoprotein (LDL) will be obtained by calculation: VLDL = TG/5; and LDL = Tchol - (VLDL + HDL). HDL: Tchol ratio will be used to evaluate the impact of treatment assignments on the lipid panel. If the PRC staff see that your lab values are abnormal, we will give you a copy of your test results and ask that you follow up with your doctor for care
Change in Blood Pressure | Up to 3 Months
  will be measured by using a Dinamap Monitor Pro 100 (GE Healthcare, Piscataway, NJ) after sitting for 5 minutes. Both systolic and diastolic pressures will be calculated as the mean value of 2 readings 5 minutes apart for each participant at every time point of assessment. If either number of your blood pressure reading is 170/110 mmHg or above, the Prevention Research Center staff will plan to escort you to the Emergency Department for care.
Change in Purchasing Behavior | Up to 3 Months
  will be tracked using the NutriSavings (www.nutrasavings.com) system which is offered to all Griffin employees. If not currently enrolled in Nutrasavings, employees will be enrolled as part of the study enrollment processes.

OTHER OUTCOMES:
Change in Physical Activity | Up to 3 Months
  Physical activity will be assessed using the International Physical Activity Questionnaire [15] Short Form to allow us to control for changes in PA that could affect outcome measures. The IPAQ is a valid and reliable tool to assess physical activity in adults. It is a more comprehensive tool containing information on weekly activities in household and yard-work activities, occupational activity, transport, leisure time physical activity and sedentary behavior.
Change in Cooking Skills | Up to 3 Months
  Participants will complete a brief survey (pre and post intervention) regarding their cooking practices and meal preparation.
Compliance | One week
  Compliance will be tracked by attendance at the weekly workshops and redemption of coupon/vouchers.
Change in Body Composition- Body Weight | Up to 3 Months
  Body composition (Body Weight) will be measured using the Tanita SC-240 Body Composition Analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Beth P Comerford, MS, Principal Investigator — Yale-Griffin Prevention Research Center; Kimberly Doughty, PhD, MPH, Study Chair — Yale-Griffin Prevention Research Center
Locations (1):
- Griffin Hospital, Derby, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Guenther PM, Dodd KW, Reedy J, Krebs-Smith SM. Most Americans eat much less than recommended amounts of fruits and vegetables. J Am Diet Assoc. 2006 Sep;106(9):1371-9. doi: 10.1016/j.jada.2006.06.002. PMID 16963342
- [Background] Benton D. Role of parents in the determination of the food preferences of children and the development of obesity. Int J Obes Relat Metab Disord. 2004 Jul;28(7):858-69. doi: 10.1038/sj.ijo.0802532. PMID 15170463
- [Background] Birch LL, Anzman-Frasca S. Learning to prefer the familiar in obesogenic environments. Nestle Nutr Workshop Ser Pediatr Program. 2011;68:187-96; discussion 196-9. doi: 10.1159/000325856. Epub 2011 Oct 3. PMID 22044900
- [Background] Fuemmeler BF, Anderson CB, Masse LC. Parent-child relationship of directly measured physical activity. Int J Behav Nutr Phys Act. 2011 Mar 8;8:17. doi: 10.1186/1479-5868-8-17. PMID 21385455
- [Background] Soler RE, Leeks KD, Razi S, Hopkins DP, Griffith M, Aten A, Chattopadhyay SK, Smith SC, Habarta N, Goetzel RZ, Pronk NP, Richling DE, Bauer DR, Buchanan LR, Florence CS, Koonin L, MacLean D, Rosenthal A, Matson Koffman D, Grizzell JV, Walker AM; Task Force on Community Preventive Services. A systematic review of selected interventions for worksite health promotion. The assessment of health risks with feedback. Am J Prev Med. 2010 Feb;38(2 Suppl):S237-62. doi: 10.1016/j.amepre.2009.10.030. PMID 20117610
- [Background] Katz DL, O'Connell M, Yeh MC, Nawaz H, Njike V, Anderson LM, Cory S, Dietz W; Task Force on Community Preventive Services. Public health strategies for preventing and controlling overweight and obesity in school and worksite settings: a report on recommendations of the Task Force on Community Preventive Services. MMWR Recomm Rep. 2005 Oct 7;54(RR-10):1-12. PMID 16261131
- [Background] Chapman LS. Meta-evaluation of worksite health promotion economic return studies: 2012 update. Am J Health Promot. 2012 Mar-Apr;26(4):TAHP1-TAHP12. doi: 10.4278/ajhp.26.4.tahp. No abstract available. PMID 22375583
- [Background] Beresford SA, Thompson B, Feng Z, Christianson A, McLerran D, Patrick DL. Seattle 5 a Day worksite program to increase fruit and vegetable consumption. Prev Med. 2001 Mar;32(3):230-8. doi: 10.1006/pmed.2000.0806. PMID 11277680
- [Background] Sorensen G, Stoddard A, Peterson K, Cohen N, Hunt MK, Stein E, Palombo R, Lederman R. Increasing fruit and vegetable consumption through worksites and families in the treatwell 5-a-day study. Am J Public Health. 1999 Jan;89(1):54-60. doi: 10.2105/ajph.89.1.54. PMID 9987465
- [Background] An R. Effectiveness of subsidies in promoting healthy food purchases and consumption: a review of field experiments. Public Health Nutr. 2013 Jul;16(7):1215-28. doi: 10.1017/S1368980012004715. Epub 2012 Nov 5. PMID 23122423
- [Background] Ball K, McNaughton SA, Le HN, Gold L, Ni Mhurchu C, Abbott G, Pollard C, Crawford D. Influence of price discounts and skill-building strategies on purchase and consumption of healthy food and beverages: outcomes of the Supermarket Healthy Eating for Life randomized controlled trial. Am J Clin Nutr. 2015 May;101(5):1055-64. doi: 10.3945/ajcn.114.096735. Epub 2015 Apr 15. PMID 25877492
- [Background] Marshall A, et al. Assessment of health-related physical activity: Results of the International Physical Activity Questionnaire Reliability and Validity Study.
- [Background] Carpenter RA, Finley C, Barlow CE. Pilot test of a behavioral skill building intervention to improve overall diet quality. J Nutr Educ Behav. 2004 Jan-Feb;36(1):20-4. doi: 10.1016/s1499-4046(06)60124-3. PMID 14756978
- [Background] Jekel J, Katz D, Elmore J. Epidemiology, Biostatistics and Preventive Medicine. 2nd ed. Philadelphia, PA: WB Saunders Company; 2001
- See also: Related Info — https://www.cdc.gov/vitalsigns/pdf/2010-08-vitalsigns.pdf